CLINICAL TRIAL: NCT02957825
Title: Surveillance of High-risk Early Postsurgical Patients for Real-time Detection of Complications Using Continuing Wireless Monitoring
Brief Title: Surveillance of High-risk Early Postsurgical Patients for Real-time Detection of Complications
Acronym: SHEPHERD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid pandemic
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Principal Investigator, B Preckel, Professor of Anesthesiology, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEPHERD
Record Dates: First submitted 2016-09-26; First posted 2016-11-08 (Estimated); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Complication, Postoperative
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Routine monitoring
- Continuous wireless monitoring (Experimental): Continuous wireless monitoring
  Interventions: Device: Continuous wireless monitoring

INTERVENTIONS:
Device: Continuous wireless monitoring — Continuous wireless monitoring of vital signs
  Arms: Continuous wireless monitoring

SUMMARY:
The aim of this study is to test the hypothesis that continuous wireless monitoring on the postsurgical ward will improve patient outcome, measured as disability-free survival at three months after surgery. Further, the investigators hypothesize that this tight control regimen decreases length of hospital stay and treatment costs in patients with complications.

DETAILED DESCRIPTION:
Every year, approximately 1,500,000 surgical procedures are performed in The Netherlands alone. After major surgery, the complication rate is conservatively estimated at 25%, with a rate of 15% for major complications. In these patients, the most important problems are a failure to timely detect developing complications and a failure to adequately rescue those patients. Currently, measurement of vital signs and standardized assessment of patient wellbeing are routinely performed intermittently for every 8-12 hours, which may lead to a failure to detect of patients with complications.

The aim of this study is to test the hypothesis that continuous wireless monitoring on the postsurgical ward will improve patient outcome, measured as disability-free survival at three months after surgery. Further, the investigators hypothesize that this tight control regimen decreases length of hospital stay and treatment costs in patients with complications.

The investigators will carry out this study as an interventional, randomized (per surgical ward), prospective, clinical trial; participating wards will be included using a stepped-wedge design.

Primary outcome is disability-free survival at three months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing acute or elective major or intermediate surgery
* American Society of Anesthesiology (ASA) score of I to IV

Exclusion Criteria:

* Inability to give written and informed consent
* Refusal to participate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 747 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Disability-free survival | 3 months
  Disability-free survival as measured by the World Health Organization Disability Assessment Schedule (WHODAS) 2.0 questionnaire

SECONDARY OUTCOMES:
Disability-free survival | 1 month
  Disability-free survival as measured by the World Health Organization Disability Assessment Schedule (WHODAS) 2.0 questionnaire
Quality of life as measured by EuroQoL questionnaire | 1 month
  EuroQol Dutch EQ-5D-5L
Quality of life as measured by EuroQoL questionnaire | 3 months
  EuroQol Dutch EQ-5D-5L
Patient Health Status | 1 month
  Short-Form Health Survey; SF-12, Dutch version
Patient Health Status | 3 months
  Short-Form Health Survey; SF-12, Dutch version
Length of hospital stay | within 30 days or until hospital discharge, whatever comes first
  Admission to discharge
In-hospital mortality | within 30 days
  Patient died during the initial hospital stay
30 day mortality | 30 days
  Did the patient die 30 days after the operation
90 day mortality | 90 days
  Did the patient die 90 days after the operation
Total number of complications | within 30 days or until hospital discharge, whatever comes first
  Total number of complications (as mentioned in the surgical discharge letter, based on the Clavien-Dindo classification) per 100 patients grated in severity
Number of patients with one or more complications (also from the surgical discharge letter) | within 30 days or until hospital discharge, whatever comes first
  Incidence of postoperative complications
Comprehensive Complication Index score (CCI) | within 30 days or until hospital discharge, whatever comes first
  The CCI is an assessment tool for a patient's overall morbidity based on the number and severity of complications
ICU admission | within 30 days or until hospital discharge, whatever comes first
  ICU admission and length of stay in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt Preckel, MD, Principal Investigator — Academic Medical Centyer Amsterdam, Anesthesiology
Locations (2):
- Netherlands (2):
  - Academic Medical Center, University of Amsterdam, Amsterdam
  - University Medical Center Utrecht (UMCU), Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Posthuma LM, Breteler MJM, Lirk PB, Nieveen van Dijkum EJ, Visscher MJ, Breel JS, Wensing CAGL, Schenk J, Vlaskamp LB, van Rossum MC, Ruurda JP, Dijkgraaf MGW, Hollmann MW, Kalkman CJ, Preckel B. Surveillance of high-risk early postsurgical patients for real-time detection of complications using wireless monitoring (SHEPHERD study): results of a randomized multicenter stepped wedge cluster trial. Front Med (Lausanne). 2024 Jan 5;10:1295499. doi: 10.3389/fmed.2023.1295499. eCollection 2023. PMID 38249988